CLINICAL TRIAL: NCT02560233
Title: Modulating Stress-Reactivity by Real-Time Multimodal Functional Neuroimaging Based Neurofeedback
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects were recruited
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Korea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GRNP_2013S1A2A2035364_1
Record Dates: First submitted 2015-08-10; First posted 2015-09-25 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Stress; Pituitary-Adrenal System
Keywords: Neurofeedback; Stress; fMRI; Real-time fMRI Neurofeedback; Anterior cingulate cortex; Hypothalamic-pituitary-adrenal axis; Cortisol; EEG; Heart rate variability; Blood pressure; Simultaneous EEG/fMRI

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingent (Experimental): Contingent RT-fMRI-NF
  Interventions: Other: Contingent RT-fMRI-NF
- Non-contingent (Sham Comparator): Sham RT-fMRI-NF
  Interventions: Other: Sham RT-fMRI-NF

INTERVENTIONS:
Other: Contingent RT-fMRI-NF — Subjects are provided with contingent RT-fMRI-NF of brain activity in the target region of interest.
  Arms: Contingent
Other: Sham RT-fMRI-NF — Subjects are provided with sham RT-fMRI-NF of brain activity of previously recorded subject.
  Arms: Non-contingent

SUMMARY:
The overall goal of the outlined study is to establish a Real-Time (RT) functional Magnetic Resonance Imaging (fMRI) Neurofeedback (NF) (RT-fMRI-NF) protocol aiming at modulating neural, endocrine, and subjective reactivity to psychosocial stress.

DETAILED DESCRIPTION:
The overall goal of the outlined study is to establish an RT-fMRI-NF protocol aiming at modulating neural, endocrine, and subjective reactivity to psychosocial stress. More specifically, the investigators pursue the following goals: a) to evaluate whether neural and subjective stress-reactivity can be modified by training volitional control over targeted brain activity by means of RT-fMRI-NF; b) to evaluate whether neuromodulation by means of RT-fMRI-NF can be used as a new way to modulate hormone-release into the periphery; and c) to evaluate whether the efficacy of neuromodulation by RT-fMRI-NF can also be reflected on EEG data as well as the autonomic nervous system (ANS) measured by heart rate variability (HRV).

ELIGIBILITY:
Inclusion Criteria:

* Sufficient spoken and written knowledge of English
* Right-handedness
* Ability to participate in study procedures

Exclusion Criteria:

* Present or past psychological or psychiatric therapy
* Major or unstable general medical conditions
* Presence of cardiovascular disease
* Current intake of any medication interfering hormonal assessments
* History of major cerebral injury
* Medical MRI contraindication

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hypothalamic-pituitary-adrenal (HPA) axis reactivity | At study day one
  Assessed via salivary cortisol
Blood oxygenation level dependent signal of the target brain region of interest | At study day one
  Blood oxygenation level dependent (BOLD) signal assessed via functional magnetic resonance imaging, expressed in relative BOLD signal intensity

SECONDARY OUTCOMES:
Psychophysiological stress reactivity - blood pressure | At study day one
  Assessed via blood pressure
Psychophysiological stress reactivity - heart rate variability | At study day one
  Assessed via heart rate variability
Psychophysiological stress reactivity - heart rate | At study day one
  Assessed via heart rate
Subjective stress reactivity | At study day one
  Assessed via Visual Analog Scale
Electrical activity of the brain | At study day one
  Assessed via electroencephalography (EEG)

OTHER OUTCOMES:
Functional connectivity | At study day one
  Connectivity of brain activity determined by fMRI signal
Feedback on adverse events during the scanner training | At study day one
  Number of subjects reporting an adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Marion Tegethoff, PD Dr., Principal Investigator — University of Basel; Jong-Hwan Lee, Prof., Principal Investigator — Korea University; Gunther Meinlschmidt, Prof. Dr., Principal Investigator — University of Basel; Ruhr-University Bochum

IPD SHARING:
Plan to Share IPD: No